CLINICAL TRIAL: NCT01626300
Title: The Effect of Milk Components on the Response to the Pneumonia Vaccine in Senior Citizens: A Randomized Placebo-controlled Clinical Trial
Brief Title: The Effect of Milk Components on the Response to the Pneumonia Vaccine in Senior Citizens
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200513884
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: The Effect of Milk Components on the Response to Pneumococcal Vaccines in the Elderly

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine if the daily use of a certain amount and type of milk component for 2 months provides a significant stimulation to the immune system and specifically increases the chances of being protected against pneumonia after the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age and a willingness to participate

Exclusion Criteria:

* • Smoking history within 10 years

  * Underlying neoplasia or immunological disease
  * Use of oral cortisone or other immunosuppressive agents
  * Current consumption of milk and milk products greater than 1 unit of milk, 1 yogurt, or 1 serving of fresh cheese a day.
  * Food faddists or those taking a non-traditional diet
  * Current consumption of dietary supplements
  * People with a known history of milk allergy
  * People with chronic renal failure
  * People with chronic inflammatory diseases taking daily doses of NSAIDs for longer than 4 weeks at the time of enrollment.
  * Previous administration of the pneumomax vaccine
  * Reduced physical activity (i.e. NYHA classes III-IV)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects > 60 years of age.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)